CLINICAL TRIAL: NCT00318045
Title: Effects of Optical Blur on Performance and Comfort of Computer Users
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vision Council of America (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: X050208014
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2006-04-25 (Estimated); Status verified 2006-04

CONDITIONS: Refractive Error
Keywords: Refractive error; Asthenopia
MeSH Terms: conditions — Refractive Errors; Asthenopia

INTERVENTIONS:
Device: Eyeglass lenses

SUMMARY:
The aim of this study is to examine the relationship between optical blur from poor refractive corrections (glasses) of workers using computers and their productivity and comfort in the workplace. We believe that improving the visual status of subjects who use computers will have a beneficial effect on productivity and visual comfort.

DETAILED DESCRIPTION:
The aim of this study is to examine the relationship between optical blur from poor refractive corrections (glasses) of workers using computers and their productivity and comfort in the workplace. We believe that improving the visual status of subjects who use computers will have a beneficial effect on productivity and visual comfort. All subjects will be required to complete a vision screening at no charge to decide if you qualify for the study. Subjects will select a frame to be worn during the period of the study. Subjects will wear either your best correction or your present prescription in the frame for a period of 1-month. This will be a double-blind study, which means that neither the subject nor your doctors will know which pair of glasses the subjects will be wearing during the parts of the study. Subjects will complete 4 hours of testing during the first period (4 weeks) then the lenses will be switched for the second period (4 weeks). During the testing, subjects will complete two tasks on a standard computer. Either the investigator or co-investigator will explain to you how to do these simple tasks. One of these tasks will involve looking at printed material and entering correct information into the computer. The other task involves finding and deleting apostrophes from a manuscript on the computer. All subjects will answer a short survey before and after these tasks to check on symptoms resulting from using the computer. Before and after each period, the subjects also will answer another survey to measure their visual functioning using these glasses.

The following periodic measurements will be made during the study: productivity and accuracy to enter a list of state populations, and a search for apostrophes (') in a document on one of the states of the U.S. These tasks will require 4 hours testing with each of the two pairs of trial glasses for two periods (each period lasts for one month). Subjects will be asked to return to the clinic for 4 hrs during the first 4-week period and for 4 more hrs during the second 4-week period. At each visit subjects will be asked if they have experienced any undesirable reactions and will complete a short survey.

Subjects will also be required to complete a short 9-question survey to determine their visual comfort before and after 1-hour of work on their own computer at your home or job during each 1-month period of the study. These short phone surveys will take less than 5-minutes to complete and will be arranged at the subject's convenience before and after the subjects are going to be working on your computer for at least 1-hr. This survey will be repeated on five occasions. Finally, 3-months after the experimental portion of the study is completed, all subjects will be required to also answer the same short 9-question survey as you work on your computer. This will also be a phone survey and will be completed on three occasions before and after 1-hr of work on their own computer at home or job.

ELIGIBILITY:
Inclusion Criteria:

* 19 yrs of age or more
* Use a computer for 1 hr per day or more
* 20/40 or better visual acuity in each eye

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2005-10; Study Completion 2006-04

PRIMARY OUTCOMES:
Visual comfort
Productivity (correct output per hour)

CONTACTS AND LOCATIONS:
Overall Officials: Kent M. Daum, O.D., Ph.D., Principal Investigator — School of Optometry, University of Alabama at Birmingham
Locations (1):
- School of Optometry, Birmingham, Alabama, United States